CLINICAL TRIAL: NCT05323149
Title: The Impact of Early Use of Tranexamic Acid in Traumatic Brain Injury Upon the Inflammatory Response and Outcome
Brief Title: Tranexamic Acid in Traumatic Brain Injury
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17101636
Record Dates: First submitted 2022-03-27; First posted 2022-04-12 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Response
MeSH Terms: interventions — Sodium Chloride; Saline Solution; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Placebo Comparator): Group C, will be received saline (loading dose of 1gm of saline 0.9%, followed by a 1gm of maintenance saline dose over 8 hours for 48 h).
  Interventions: Other: Saline
- Group T (Experimental): Group T, will be received TXA (loading dose of 1gm of TXA, followed by a 1gm of maintenance dose over 8 hours for 48 h).
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Other: Saline — Giving saline (loading dose of 1gm of saline 0.9%, followed by a 1gm of maintenance saline dose over 8 hours for 48 h).
  Other Names: Normal saline
  Arms: Group C
Drug: Tranexamic acid — Giving TXA (loading dose of 1gm of TXA, followed by a 1gm of maintenance dose over 8 hours for 48 h).
  Other Names: Cyclokapron
  Arms: Group T

SUMMARY:
In this study, our aim is to investigate the role of tranexamic acid for modulating the inflammation in patients with traumatic brain injury (TBI).

DETAILED DESCRIPTION:
This is double-blind trial, where group T will be received TXA, where group C will be received saline placebo.

In emergency room (ER), trauma patients will be assessed and managed according to our local hospital protocol. After the initial resuscitation of patients. The selection was done according to the inclusion criteria. Baseline investigations

1. C-reactive protein (CRP), interleukin -6(IL-6), C-reactive protein/Albumin ratio (CAR), complete blood count (CBC) for neutrophil lymphocyte ratio (NLR), platelet lymphocyte ratio (PLR).
2. Prothrombin concentration (PC), prothrombin time (PT), activated partial thromboplastin time (aPTT), and INR.

Group T, will be received TXA (loading dose of 1gm of TXA, followed by a 1gm of maintenance dose over 8 hours for 48 h). Group C, will be received saline (loading dose of 1gm of saline 0.9%, followed by a 1gm of maintenance saline dose over 8 hours for 48 h) to monitor the post-interventional inflammatory response (CBC for NLR, PLR), CRP, IL-6, C-reactive protein/Albumin ratio (CAR), hemostasis (PC, PT, activated PTT, and international normalized ratio (INR)) and short-term outcome. Conscious level will be assessed by Glasgow come scale (GCS), delirium by Richmond Agitation-Sedation Scale (RASS score) and hemodynamics will be continuously monitored. Patients will be monitored and managed in intermediate or intensive care unit. Adverse effects and complications will be recorded and managed.

ELIGIBILITY:
Inclusion Criteria:

* Isolated traumatic brain injury patients (mild or moderate cases)
* GCS > 8
* non penetrating TBI in 8 hours onset
* Age ≥ 18 years

Exclusion Criteria:

* Patient in cardiac arrest
* Patients with coagulopathies
* Renal failure patients
* pregnancy
* Patient refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2027-09-10 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with decreased the inflammatory response | 48 hours post-interventional (either placebo or TXA)
  Percentage of patients with decreased the inflammatory response, as assessed by NLR measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided